CLINICAL TRIAL: NCT04081662
Title: Examining the Efficacy of Acceptance and Commitment Therapy (ACT) Microinterventions for Distressed First-Generation College Students
Acronym: CompACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0819; Biostat & Med (Other: UW, Madison); A538900 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison)
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Psychological Distress; Self-Assessment; Mood Change
Keywords: Acceptance and commitment therapy; Micro-intervention; Mobile intervention

STUDY DESIGN:
Intervention Model Description: This study uses a design known as a microrandomized trial. Whereas a multi-arm trial randomizes a subject to an intervention group only once at the start of the study, a microrandomized trial repeatedly randomizes a subject to an intervention group throughout the study. In addition to an overall effect of an intervention on proximal outcomes, a microrandomized trial allows one to determine if the effect is modified by momentary factors (e.g., current mood, day of the week, day in the study).
  For the present study, every subject has a equal chance of being assigned to one of two intervention groups at each of 84 time points (2 daily x 42 days). At each time point, the two intervention groups are to either receive a prompt based on Acceptance and Commitment Therapy (ACT) or not receive such a prompt. Regardless of the assigned group, subjects are asked to assess their mood, stress, and activity at every time point prior to assignment to intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- compACT Intervention (Experimental): At every time-point of the study, participants will complete self-reports of stress, (as measured by the PSS-4) distress (as measured by the PHQ-2), and activity through the mobile app Lorevimo. After completing these assessments, participants will be randomly assigned to either receive one additional ACT-based microintervention question or receive no additional question.
  The microintervention will consist of one of 84 prompts that aim to target one of 6 processes targeted in ACT (contacting the present moment, defusion, acceptance, self-as-context, values, and committed action).
  The ACT-based questions were developed by the research team as a unique intervention for the current study. They are based upon core themes of acceptance and commitment therapy: engagement, awareness, and openness.
  Interventions: Behavioral: compACT Intervention

INTERVENTIONS:
Behavioral: compACT Intervention — The mobile intervention in this study consists of two components: 1) self-monitoring and 2) an ACT-based microintervention.
  Self-monitoring: twice daily, participants will complete self-reports of distress, depressive symptoms, and activity through the mobile app Lorevimo.
  Microintervention: The microintervention will consist of one of 84 prompts that aim to target one of 6 processes targeted in ACT (contacting the present moment, defusion, acceptance, self-as-context, values, and committed action). At each time-point, participants have a 50% chance of receiving a microintervention question along with the daily self-monitoring assessments.

SUMMARY:
This research study aims to evaluate the feasibility, safety, and effectiveness of a micro-randomized acceptance and commitment therapy-based (ACT-based) intervention that is delivered to distressed first-generation college students.

DETAILED DESCRIPTION:
The transition to college is associated with a number of changes in health behaviors and mental health functioning, with 50% of college students meeting criteria for a psychiatric disorder. In particular, first-generation college students may be at particular risk for increased stress and mental health difficulties. The development of effective psychotherapeutic interventions is essential in providing adequate care to young adults during the transitional years of college. Delivery of these interventions via acceptable and feasible modalities for this population is also of utmost importance so that utilization and engagement are prioritized. Brief interventions have been a point of emphasis in recent years from the perspective of patient and provider efficiency, as well as many studies indicating effectiveness of brief interventions in creating and sustaining clinical levels of change.

The current study seeks to evaluate the effectiveness of brief interventions delivered via a smartphone app, or "microinterventions", based in Acceptance and Commitment Therapy (ACT). ACT is a cognitive-behavioral therapy that seeks to promote psychological flexibility. ACT is transdiagnostic, meaning that it is designed to target human suffering, rather than a particular psychological or physical disorder. ACT targets experiential avoidance, which is the inability or unwillingness to make contact with painful experiences (e.g., thoughts, emotions, memories. Avoidance provides short-term relief, but exacerbates the long-term experience of the avoided stimulus in terms of intensity and duration. The microintervention in this study will consist of one of 84 prompts that aim to target one of 6 processes targeted in ACT. For example, one prompt is "Do your current actions align with what matters most to you?" Delivery of these prompts (e.g., whether and when to deliver which prompt) is randomized to allow for secondary analyses of optimal delivery of the microintervention in addition to primary analyses of its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide informed consent.
2. Willing to comply with all study procedures and be available for the duration of the study.
3. Individuals 18-19 years of age.
4. Individuals who are full-time freshman or sophomore students at the University of Wisconsin-Madison.
5. Fluent in written English.
6. Has access to a smartphone.
7. First-generation college student.
8. Significant subjective distress (endorses distress on at least 4 out of the past 7 days that interfered with functioning in screening survey).

Exclusion Criteria:

1. Expected life expectancy <6 months.
2. Use of investigational drugs, biologics, or devices within 30 days prior to randomization.
3. Not suitable for study participation due to other reasons at the discretion of the investigators.

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of the ACT micro-intervention: percentage adherence to PHQ-2, PSS-4, and activity prompts | Day 1 - day 43
  The feasibility of the microintervention will be assessed by Adherence to prompts (defined as a response to at least 50% completion of prompt items per day). If subjects adhere to prompts over 60% of the days of the intervention period on average, the intervention will be considered feasible. The prompts considered will be the 2 questions from the PHQ-2, the 4 questions from the PSS-4, and the 4 questions from the activity assessment.
Safety of ACT micro-intervention: Change in Patient Health Questionnaire 9 (PHQ-9) | Baseline, 3 months and 6 months post intervention
  The analysis will look at the change in proportion of individuals who meet criteria for minor or major depression on the PHQ-9 between study start (measure taken at baseline assessment) to study end (measure taken at 6-month follow-up assessment).
  The Patient Health Questionnaire 9 (PHQ-9) is a multipurpose scale for screening, diagnosing, monitoring and measuring the severity of depression. PHQ-9 will reflect the effect of intervention on the severity of depression. The PHQ-9 scores correlates with the depression severity as follows:
  5 to 9- Minimal symptoms 10 to 14- Minor depression 15 to 19 Major depression, moderately severe >20 Major depression, severe
Effectiveness of the ACT micro-intervention: proximal changes in mood outcomes as a result of intervention as indicated by self-reported activity of participant | Days 1-43
  The effectiveness of the ACT micro-intervention will be assessed by looking at the responses to the activity assessment in relation to whether or not a participant received a micro-intervention at the prior time-point. The activity questions of interest are as follows:
  1. Since you [woke this morning or last logged your symptoms], how much energy was consumed by trying to get rid of unwanted feelings, thoughts, or other internal experiences (example: suppressing, distracting, avoiding)?
  2. Since you [woke this morning or last logged your symptoms], how much energy was consumed by pursuing your values (example: making choices that align with who you want to be or who/what matters)?
  Both questions are answered using a scale of 0-6, where 0 = "none" and 6 = "all of my energy."

SECONDARY OUTCOMES:
Proximal changes in mood outcomes as a result of intervention: The Perceived Stress Scale (PSS-4) score | Days 1-43
  The effectiveness of the ACT micro-intervention will be assessed by looking at the PSS-4 score in relation to whether or not a participant received a micro-intervention at the prior time-point.
  The Perceived Stress Scale (PSS-4) consists of four questions, each answered using a scale of 0-4. The total PSS-4 score ranges from 0-16. A higher score indicates a higher degree and/or longer duration of perceived stress.
Proximal changes in mood outcomes as a result of intervention: Patient Health Questionnaire-2 (PHQ-2) score | Days 1-43
  The effectiveness of the ACT micro-intervention will be assessed by looking at PHQ-2 score in relation to whether or not a participant received a micro-intervention at the prior time-point. The PHQ-2 consists of the first two questions of the Patient Health Questionnaire-9 (PHQ-9) and asks about the frequency of depressed mood and anhedonia over the past two weeks. Each question is answered on a scale of 0-3 as follows:
  0 = Not at all
  1. = Several days
  2. = More than half the days
  3. = Nearly every day
  The PHQ-2 score ranges from 0-6, with a score of 0-2 being negative for potential major depressive disorder and a score of 3 or more being positive for potential major depressive disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas EBK, Sagorac Gruichich T, Maronge JM, Hoel S, Victory A, Stowe ZN, Cochran A. Mobile Acceptance and Commitment Therapy With Distressed First-Generation College Students: Microrandomized Trial. JMIR Ment Health. 2023 May 15;10:e43065. doi: 10.2196/43065. PMID 37184896
- [Derived] Kroska EB, Hoel S, Victory A, Murphy SA, McInnis MG, Stowe ZN, Cochran A. Optimizing an Acceptance and Commitment Therapy Microintervention Via a Mobile App With Two Cohorts: Protocol for Micro-Randomized Trials. JMIR Res Protoc. 2020 Sep 23;9(9):e17086. doi: 10.2196/17086. PMID 32965227